CLINICAL TRIAL: NCT06635850
Title: A Phase 2, Randomized, Placebo-Controlled Trial to Assess the Efficacy and Safety of Mosliciguat in Participants With Pulmonary Hypertension Associated With Interstitial Lung Disease
Brief Title: A Study of Mosliciguat in PH-ILD
Acronym: PHocus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmovant, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-2301-201
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease; Lung Diseases; Vascular Diseases; Cardiovascular Diseases; Fibrosis
Keywords: PH; ILD; 6 Minute Walk Test; mosliciguat
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial; Lung Diseases; Vascular Diseases; Cardiovascular Diseases; Fibrosis | interventions — Dry Powder Inhalers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Mosliciguat (Active Comparator): Participants will be randomized to receive inhaled mosliciguat or placebo daily for 24 weeks
  Interventions: Drug: Mosliciguat; Device: Dry Powder Inhaler
- Matched Placebo (Placebo Comparator): Participants will be randomized to receive inhaled mosliciguat or placebo daily for 24 weeks
  Interventions: Device: Dry Powder Inhaler; Drug: Placebo
- Extension (Experimental): After Week 24, all participants may receive mosliciguat through an Extension period
  Interventions: Drug: Mosliciguat; Device: Dry Powder Inhaler

INTERVENTIONS:
Drug: Mosliciguat — Dose level 1, 2, or 3 for inhalation
  Arms: Extension; Mosliciguat
Device: Dry Powder Inhaler — Dry powder inhaler for mosliciguat or placebo delivery
Drug: Placebo — Matching placebo for inhalation
  Arms: Matched Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, multi-center clinical study to evaluate the safety and efficacy of inhaled mosliciguat in participants with pulmonary hypertension associated with interstitial lung disease (PH-ILD).

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled study with an extension.

The study consists of 2 periods: a blinded placebo-controlled period (24 weeks) and an extension (beyond 24 weeks).

Participants will be randomized to receive mosliciguat or placebo in the 24-week double-blind treatment period.

All participants who complete the 24-week double-blind period may continue to participate in the extension period where all participants will receive mosliciguat.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to provide informed consent
* Participants with diagnosis of Interstitial Lung Disease (ILD). Diagnosis will be confirmed by a high-resolution computerized tomography (HR-CT) scan showing diffuse parenchymal disease. Eligible diagnosed diseases include:

  1. Idiopathic interstitial pneumonia (IIP)
  2. Chronic hypersensitivity pneumonitis
  3. ILD associated with connective tissue disease (CTD) with a forced vital capacity (FVC) < 70% of predicted
* Confirmed pulmonary hypertension (PH) by right heart catheterization (RHC).
* Ability to perform 6MWD ≥100 meters.

Exclusion Criteria:

* Diagnosis of PH Group 1 (eg. pulmonary arterial hypertension), Group 2 (related to left-heart dysfunction), Group 4 (eg, chronic thromboembolic pulmonary hypertension), or Group 5 (eg, unclassified).
* Exacerbation of underlying lung disease within 28 days prior to randomization.
* Initiation of pulmonary rehabilitation within 28 days prior to randomization.
* Receiving >10 L/min of oxygen supplementation by any mode of delivery at rest at Baseline.
* History or intolerance to or lack of efficacy with mosliciguat or sGC stimulators or activators.
* Receipt of investigational, or experimental therapy within 42 days OR 5 half-lives prior to randomization.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 16 in Pulmonary Vascular Resistance (PVR) | Baseline, Week 16
  PVR evaluated using right heart catheterization (RHC).

SECONDARY OUTCOMES:
Change from Baseline to Week 16 in Distance Achieved on the Six-Minute Walk Test (6MWT) | Baseline, Week 16
  The 6MWT measures the distance a participant is able to walk quickly on a flat, hard surface in a period of 6 minutes.
Change from Baseline to Week 16 in N-terminal pro-brain natriuretic peptide (NT-proBNP) | Baseline, Week 16
  The NT-proBNP serum concentration is a useful biomarker associated with changes in right heart morphology and function. NT-proBNP serum concentration will be assessed to compare the severity of heart failure at Baseline and Week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Ubaldo Martin, MD, Study Director — Pulmovant, Inc.
Locations (18):
- United States (18):
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California Davis School of Medicine, Sacramento, California
  - Harbor-UCLA Medical Center - Torrance, Torrance, California
  - Florida Lung, Asthma & Sleep Specialists/Clinical Research Specialists, LLC, Celebration, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - Duke University Health System - Duke Clinic, Durham, North Carolina
  - PulmonIx, Greensboro, North Carolina
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Summit Health, Bend, Oregon
  - Lewis Katz School of Medicine, Philadelphia, Pennsylvania
  - Brown Medicine, East Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Lung Center, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah

REFERENCES:
- See also: Related Info — https://phocusstudy.com/